CLINICAL TRIAL: NCT04900831
Title: Validation of Beat-to-beat Wavefront Direction Using Omnipolar Mapping
Acronym: ATOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 19HH5064
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Atrial Flutter Typical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Diagnostic Test: Omnipolar Eletroanatomical mapping

INTERVENTIONS:
Diagnostic Test: Omnipolar Eletroanatomical mapping — Analyse intracardiac EGMs collected with the HD Grid catheter (Abbott, Chicago, IL) during routine Atrial Flutter ablation using the Omnipolar algorithm.

SUMMARY:
To validate omnipolar mapping in a well-described circuit within the heart (Atrial Flutter) and compare it with the gold standard of Local Activation Time (LAT) mapping during routine, clinically indicated procedures of Atrial Flutter ablation. A conventional, LAT map will be created during the procedure, prior to treatment, to guide the procedure. A repeat map will be performed after ablation during the procedure. The investigators will export the map files for off-line analysis with the omnipolar software.

DETAILED DESCRIPTION:
Electroanatomical mapping of the chambers of the heart has revolutionised the way physicians treat heart rhythm disorders. However, there still are technical limitations that prevent us from gathering information that could be used to understand and treat these abnormal circuits in more detail.

The gold standard technique in creating electrical maps of the heart in stable circuits is the Local Activation Time (LAT) map. This map is formed by using a stable electrical point (one of the electrode catheters within the heart - plastic tubes with metallic sensors at the end) as a zero point and then collecting electrical data from around the heart based on timings off of that point. This data is then loaded on a licenced software that creates the map. These maps are very useful in creating electrical maps of the heart in relatively stable electrical circuits and can give us information on how the electrical current travels through the heart tissue. These are widely used in guiding ablation by helping us locate areas to ablate (apply local radiofrequency and burn part of the circuit, deactivating it).

In more unstable circuits, such as in Atrial Fibrillation (chaotic electrical activity at the top left chamber of the heart), there are a lot of limitations of this technology as the electrical current changes from heart beat to heart beat and there is no stable zero point In the circuit to "anchor" the map in time. In these situations real-time map creation with local electrical currents would be ideal as it would help us see the direction the electrical wave front travels in real time. Our current electrical catheters have certain limitations which mainly have to do with difficulty in local electrical discrimination and detection of the orientation of the electrical current in real time.

The Advisor HD Grid catheter by Abbott UK can overcome this hurdle. It has a special electrode configuration (4 by 4) that creates 9 distinct anatomical spaces within the catheter grid that can "triangulate" micro current direction in real time (omnipolar mapping). This will greatly enhance our ability to quickly detect electrical wave fronts in unstable circuits such as Atrial Fibrillation which will lead to better understanding of the arrhythmia and identify targets for treatment quickly and efficiently.

The investigators aim to first validate the robustness of omnipolar mapping in a well-described, stable circuit such as Atrial Flutter, and compare it to the gold standard of LAT mapping. This will then help pave the way for use of this technology in more complex circuits, such as Atrial Fibrillation.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients on the waiting list for radiofrequency ablation of Atrial Flutter at the Hammersmith Hospital, Imperial College Healthcare NHS Trust.

1. Suitable candidate for catheter mapping/ablation of arrhythmias.
2. Eighteen (18) to eighty-five (85) years of age.
3. Body Mass Index (BMI) <40 (Wt. in Kgs / Ht. in cm).
4. Signed Informed Consent.

Exclusion Criteria:

1. Severe cerebrovascular disease
2. Moderate to severe renal impairment (eGFR<30 ml/min/1.73m2)
3. Active gastrointestinal bleeding.
4. Active infection or fever.
5. Short life expectancy.
6. Significant anaemia.
7. Severe uncontrolled systemic hypertension.
8. Severe electrolyte imbalance.
9. Ejection fraction <35%.
10. Congestive heart failure (NYHA IV).
11. Unstable angina requiring emergent PTCA (percutaneous transluminal coronary angioplasty) or CABG (Coronary Artery Bypass Grafting).
12. Recent myocardial infarction.
13. Bleeding or clotting disorders.
14. Uncontrolled diabetes.
15. Inability to receive IV or oral Anticoagulants.
16. Unable to give informed consent (these patients would not be recruited).
17. Previous catheter or surgical ablation treatment for Atrial Fibrillation.
18. Previous catheter ablation treatment for Atrial Flutter.
19. Pregnancy (urinary pregnancy test will be offered on the day of the procedure for all women of reproductive age)
20. Drug and/or alcohol abuse.
21. Patients who have participated in another study of an investigational medicinal product in the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent Atrial Flutter that have been listed on a clinical basis to have a Cavotricuspid Isthmus ablation (Atrial Flutter Ablation).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Omnipolar real time wavefront direction is non inferior to LAT map. | 1 year
  Maps will be compared post EP Study.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.